CLINICAL TRIAL: NCT00476788
Title: Fast Track Continuous Subcutaneous Insulin Infusion (CSII) in Children With Newly Diagnosed Type 1 Diabetes Mellitus: An Evaluation of a Novel CSII Device in the Immediate Period Following Diagnosis of Type 1 Diabetes (T1DM)
Brief Title: Fast Track CSII Using a Novel Device in Young Children With Newly Diagnosed T1DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michael Stalvey, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X060928006
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Results first posted 2011-01-24 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: pediatrics; CSII; diabetes; C-peptide; adverse events
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omnipod Device (Experimental): Patients will be placed on an Omnipod insulin pump
  Interventions: Device: Omnipod Insulin Management System

INTERVENTIONS:
Device: Omnipod Insulin Management System — Initiation of insulin pump therapy within three months of the diagnosis of type 1 diabetes mellitus
  Other Names: Tubeless insulin pump

SUMMARY:
This study evaluates early initiation of continuous subcutaneous insulin infusion (CSII) therapy in young children using a novel delivery method in the form of a self-contained, lightweight, and disposable insulin pump unit controlled with a wireless handheld device. The outcomes of interest are the feasibility and potential metabolic benefits of this approach. We anticipate that the initiation of this CSII device in the immediate post-diagnosis period in this population will result in good glycemic control and greater parental satisfaction when compared to intensive insulin injection therapy.

DETAILED DESCRIPTION:
The incidence of type 1 diabetes (T1DM) is on the rise worldwide, especially in children younger than six years of age. Glycemic control using multiple daily injection (MDI) therapy can be difficult to achieve and maintain in the very young, especially in the immediate post-diagnosis period. This study evaluates early initiation of continuous subcutaneous insulin infusion (CSII) therapy in young children using a novel delivery method in the form of a self-contained, lightweight, and disposable insulin pump unit controlled with a wireless handheld device. The outcomes of interest are the feasibility, safety, and potential metabolic benefits of this approach. We will recruit 14 pediatric patients, aged one to ten years, from a pool of all children newly diagnosed with T1DM admitted to the Children's Hospital of Alabama to use the pump.General diabetes education and CSII-specific training will take place in a series of outpatient sessions with the PI and study nurse. Pump therapy will be initiated within two months of diagnosis providing that all requisite education and training has been successfully completed. Data will be collected for both study group and control group patients for six months via phone calls and monthly clinic visits. Areas which will be evaluated include glycemic control, residual endogenous insulin secretion, frequency of severe adverse events, parental distress, insulin needs, and physical growth. While initiating CSII in the immediate post-diagnosis period in this population may be initially time-intensive, it is anticipated that it will ultimately become time-saving because of the greater ease in blood sugar management.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1 through 10 years of age
* Patients present to the Children's Hospital of Alabama with a new diagnosis of type 1 diabetes
* Patients may be admitted to the inpatient unit
* OR from the ER
* OR or from an outside facility to Children's Hospital
* Or seen in our outpatient clinic for the first time having been diagnosed at an outside facility
* If patients are recruited from the outside facility in our outpatient clinic, the diagnosis must have been made within two weeks of the visit. Twenty patients and twenty control subjects will be recruited over a six-month period.

Exclusion Criteria:

* Patients with diabetes due to other causes (neonatal diabetes, pancreatitis, cystic fibrosis, etc.)
* Patients will younger than 2 years of age
* Patients older than 8 years of age
* Lack any presence of other systemic disease(s), such as neoplastic disease or renal failure.
* Patients must have adequate parental support and stable home environment (e.g. children in foster care or with a history of suspected abuse or neglect would be excluded).

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2007-04; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine C Moreland, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Children's Hospital, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omnipod Device
Started | 14
Completed | 11
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Omnipod Device
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.275 (2.875)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Secondary Outcome: Number of Reported Adverse Events
Description: adverse events are defined as a change from baseline
Time Frame: 6.9 months (average)
Measure: Number; unit: events
Arm/Group | Omnipod Device
Number analyzed (Participants) | 11
events | 0

2. Primary Outcome: Mean Glycated Hemoglobin (A1c)
Description: Measure of glycemic control (A1c) over preceding 8 weeks. Normal for a patient between ages 1 and 10 years would be 7.0-8.5%.
Time Frame: 6.9 months (average)
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Omnipod Device
Number analyzed (Participants) | 11
percentage of glycated hemoglobin | 7.6 (1.0)

ADVERSE EVENTS:
Arm/Group | Omnipod Device
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No